CLINICAL TRIAL: NCT03413956
Title: A Multi-centre Real-world Non-interventional Observational Study to Explore Clinical Characteristics of the Chinese Patients With T1 Non-small Cell Lung Cancer Complicated With Lymph Metastases
Brief Title: An Observational Study to Explore Clinical Characteristics of the Patients With T1 Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Feng Jiang, Associate professor, Jiangsu Cancer Institute & Hospital
Other Study IDs: JS-LC-01
Record Dates: First submitted 2018-01-15; First posted 2018-01-29 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Chinese; T1 non-small cell lung cancer; Lymph metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients with lymph metastases: Pathologically diagnosed patients with T1 non-small cell lung cancer complicated with lymph metastases after surgeries
  Interventions: Procedure: Surgeries

INTERVENTIONS:
Procedure: Surgeries — Surgeries

SUMMARY:
The real-world observational study was designed to explore the odd factors of lymph metastases in the patients with T1 non-small cell lung cancer, the effects of clinical characteristics on lymph metastases, and compare the differences in lymph metastases in the subgroups.

DETAILED DESCRIPTION:
The trial is a multi-centre, real-world non-interventional observational study. In the study, the patients with T1 non-small cell lung cancer enrolled in clinics from 2015 to 2017 were included via a retrospectively review method and the study data on patient demographic/tumor biological characteristics, and clinical treatments were collected to explore the clinical odd factors of lymph metastases, evaluate the effects of clinical characteristics on lymph metastases, and compare the differences in lymph metastases in the subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received surgeries from 2015 to 2017;
* Pathologically diagnosed patients with T1 non-small cell lung cancer;

Exclusion Criteria:

- Patients with tumor treatments (including chemotherapies, radiotherapies, biological therapies, intervention therapies)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The eligible subjects are the Chinese T1 patients with non-small cell lung cancer complicated with lymph metastases
Sampling Method: Non-Probability Sample
Enrollment: 10885 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Percentage of the patients with lymph metastases | 2015 - 2017
  Percentages of the patients with lymph metastases categorised by patient demographic and tumor biological characteristics

SECONDARY OUTCOMES:
Percentages of N0/N1/N2/N3 patients | 2015 - 2017
  Percentages of N0/N1/N2/N3 patients in the target population

OTHER OUTCOMES:
Percentage of N2 patients with lymph nodes | 2015 - 2017
  Percentages of N2 patients with lymph nodes in N2 population
Percentage of patients with lymph metastases categorised by tumor baseline characteristics | 2015 - 2017
  Percentage of patients with lymph metastases categorised by tumor baseline characteristics
Number of lymph nodes in N2 patients | 2015 - 2017
  Number of lymph nodes in N2 patients categorised by tumor baseline characteristics
Percentage of patients with N2 skip metastases | 2015 - 2017
  Percentage of patients with N2 skip metastases categorised by tumor baseline characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Lin Xu, Principal Investigator — Jiangsu Cancer Institute and Hospital
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China People's Liberation Army Hospital, Beijing, Beijing Municipality
  - Henan cancer hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College, Huaxi Technology University, Wuhan, Hubei
  - Jiangsu Cancer Institute and Hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - First Hospital Affiliated to Medical College, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No